CLINICAL TRIAL: NCT03013166
Title: Resource Use and Clinical Outcomes in Patients With Adrenal Insufficiency Prescribed Either an Immediate Release or Modified Release Hydrocortisone Formulation or Prednisolone: A THIN (The Health Improvement Network) Database Study
Brief Title: THIN Database Study: Resource Use and Outcomes in Patients With Adrenal Insufficiency Prescribed Hydrocortisone: Immediate, or Modified Release, or Prednisolone
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SHP617-701
Record Dates: First submitted 2016-10-20; First posted 2017-01-06 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Cohort 1: IR hydrocortisone
  Interventions: Other: Corticosteroid medication
- Cohort 2: IR prednisolone
  Interventions: Other: Corticosteroid medication
- Cohort 3: MR hydrocortisone
  Interventions: Other: Corticosteroid medication
- Cohort 4: IR to MR hydrocortisone
  Interventions: Other: Corticosteroid medication

INTERVENTIONS:
Other: Corticosteroid medication — Patients will be grouped into Cohort 1 (IR hydrocortisone), cohort 2 (IR prednisolone), cohort 3 (MR hydrocortisone), or cohort 4 (IR to MR hydrocortisone) depending on which oral corticosteroid medications were received during the observation period.

SUMMARY:
To describe clinical outcomes and both primary and secondary care health care resource use in patients who have been prescribed either immediate-release (IR) hydrocortisone or modified-release (MR) hydrocortisone or prednisolone in the UK.

ELIGIBILITY:
Inclusion Criteria:

1. Cohort 1 (IR hydrocortisone): All patients with a Read code for AI and a prescription of IR hydrocortisone between 2010 and data extraction but no prescription for MR hydrocortisone at any time during this period, and no earlier prescription for IR prednisolone during this period
2. Cohort 2 (IR prednisolone): All patients with a Read code for AI and a prescription of IR prednisolone between 2010 and data extraction but no prescription for MR prednisolone at any time during this period, and no earlier prescription for IR prednisolone during this period
3. Cohort 3a (MR Hydrocortisone): All patients with a Read code for AI and a prescription of MR hydrocortisone between 2010 and data extraction
4. Cohort 3b (IR to MR hydrocortisone): A sub-set of patients from cohort 3a, who have switched from IR to MR hydrocortisone.
5. A list of pre-defined READ codes will be used to identify all patients with primary or secondary AI or CAH in the THIN database.

Exclusion Criteria:

1)Patients who have not received a prescription of hydrocortisone or prednisolone in the past five years will be excluded as the aim of the study is to describe recent experience.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients in the THIN database who have a Read code for AI and have been prescribed either IR hydrocortisone or prednisolone or MR hydrocortisone (plenadren) between 2010 and the date of data extraction will be included
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Primary care resource use per year in all patients as measured by using number of primary care contacts | 4 months
Primary care resource use per year in all patients as measured by number of referrals to secondary care (by specialty) | 4 months
Primary care resource use per year in all patients as measured by number of sick notes issues | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda